CLINICAL TRIAL: NCT01402856
Title: Teenage Driving Safety Study: An Emergency Medicine-Trauma Collaborative Study
Status: Completed | Type: Observational
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Marna Rayl Greenberg, Director of EM Research, Lehigh Valley Hospital
Other Study IDs: 1-20071204
Record Dates: First submitted 2011-07-08; First posted 2011-07-26 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Trauma
Keywords: Prevention; Adolescent; Trauma; Driving
MeSH Terms: conditions — Wounds and Injuries | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Southern Lehigh HS, PA School District: This school will not receive the education, yet, will be surveyed, quizzed and observed at the same time.
  Interventions: Other: Education
- Bethlehem HS, PA Area School District: Freedom & Liberty HS's in Bethlehem, PA will serve as the study's control group.
- Phillipsburg HS, NJ Area School District: This school will not receive the education, yet, will be surveyed, quizzed and observed at the same time.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — An educational program targeting HS students on the risks of distracted driving that was 60-min long & utilized: a 5-10 min DVD on a teenager's real-life experience of the devastating effects of distracted driving, other videos placing the viewer in the driver's seat, power point presentations of state and national statistics related to seat belt usage, mortality, and substance use, overview of state laws, demonstrations of the physics of an accident, & interactive games simulating distracted driving.
  Groups: Phillipsburg HS, NJ Area School District; Southern Lehigh HS, PA School District

SUMMARY:
Teenage driving safety continues to be a major public health issue. Two factors have been found to contribute to a higher teenage driving accident rate than adults: lack of driving experience, and risky behaviors. Insufficient driving experience puts teenagers at a disadvantage in detecting and responding to hazards while driving. Factors contributing to distracted driving (a diversion in the driver's attention from the road) may include: talking or text messaging on a cell phone, applying makeup, having multiple passengers, listening to loud music, eating/drinking, smoking or reading while driving.

This is a prospective study designed to evaluate the effect of an educational program on the risks associated with distracted driving for teenage drivers. The researchers will compare cell phone usage behaviors in Pennsylvania, where no cell phone laws are in place, and New Jersey, where cell phone laws exist, and will educate the beginner driver on the potential dangers associated with driving without a seat belt, substance use, and participating in distracting driving behaviors. Knowledge of state laws will also be assessed.

Objectives

1. Educate participants on the potential dangers of distracted driving.
2. Evaluate the impact of the educational program on teenage distracted driving behaviors by obtaining and analyzing information from student surveys, state law quizzes, and anonymous observation, pre, post, and delayed post education.
3. Quantify distracted driving behavior in teenage driver's attending local area high schools by obtaining and analyzing information from student surveys, state law quizzes, and anonymous observation, pre, post, and delayed post education.
4. Qualify distracted driving behavior in teenage driver's attending local area high schools by obtaining and analyzing information from student surveys, anonymous observation, and anonymous voicemails, text messages, and/or emails pre, post, and delayed post education.

Qualify distracted driving behavior in adults through anonymous observations near local area high schools.

6. Compare teenage driving behaviors as reported and observed between Pennsylvania and New Jersey.

7. Compare seat belt usage, driving behaviors, and substance use in the study population to the state and national averages pre and post education.

8. Compare averages of student's knowledge of state driving laws pre and post education.

DETAILED DESCRIPTION:
Within the 2007-2008 school year, Phillipsburg High School in Phillipsburg, New Jersey, and Southern Lehigh High School in Center Valley, Pennsylvania have agreed to take part in an educational program targeting high school students on the risks associated with distracted driving behaviors. The educational program will be approximately 60-minutes in length utilizing education material including but not limited to: a 5-10 minute DVD illustrating a teenager's real-life experience of the devastating effects of distracted driving, other videos placing the viewer in the driver's seat, power point presentations of state and national statistics related to seat belt usage, mortality, and substance use, overview of state laws, demonstrations relating to the physics of an accident, and interactive games simulating driving while distracted.

As part of the educational program, teachers will be asked to distribute an anonymous survey and a state law quiz to the students. The teachers will be provided with scripted material to use for describing the purpose of the activity and for instructing the students how to fill out the survey and state law quiz. This data will be obtained at three different time intervals (pre education, post education, and delayed post education) and will assess driving and distracted driving behaviors such as seat belt use, cell phone use, audio habits, eating while driving, substance use, personal hygiene habits, frequency and number of passengers, and knowledge of state laws.

During the educational program, students will be given an anonymous research phone number and/or email address for which they will be encouraged to leave any voicemails, text messages, and/or emails with experiences they feel are important to teenage driving. Qualitative data obtained from any anonymous communication will be received by a non-study team member, and will be sanitized of all caller numbers or identifiers.

In addition to the educational program, study team members will anonymously observe student and adult drivers pulling into and out of school parking lots, or around school property, in order to qualify their driving behaviors. Observed behaviors of students and adults will be compared for any similarities. Observers will record seat belt use, number or passengers in cars and any other witnessed distracted driving behaviors. Observations will be anonymous and will not take place on school property. Student observations will take place pre, post, and delayed post the education session. Adult observations will occur one time, independent of student observations, as the adults will not be receiving the educational intervention provided by the study. Freedom and Liberty High Schools in Bethlehem, Pennsylvania, will be utilized as the control group for this study. These schools will not receive the education, however, will be surveyed, quizzed and observed at the same time intervals as the study group.

ELIGIBILITY:
Inclusion Criteria:

1. Teenagers perceived to be students driving near school property.
2. Teenagers perceived to be of driving age.
3. Teens in 10th, 11th, and 12th grades attending Phillipsburg, Southern Lehigh, Freedom and Liberty High Schools.
4. Any driver driving near school property, which is perceived to be older than of high school age.

Exclusion Criteria:

1. Teenagers perceived as non-attendees of the nearby school.
2. Teenagers perceived not to be of driving age.
3. Teens not in 10th, 11th, and 12th grades, or not attending Phillipsburg, Southern Lehigh, Freedom and Liberty High Schools.
4. Any driver who does not meet the above criteria.

   -

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Students in the tenth, eleventh, and twelfth grades
Sampling Method: Non-Probability Sample
Enrollment: 3750 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in distracted driving behavior at one year | up to one year
  distracted driving behaviors will be quantified by anonymous observations, state law quiz results, anonymous observations, anonymous text messages/emails/voicemails pre-, post and delayed post education

CONTACTS AND LOCATIONS:
Overall Officials: Gavin C Barr, Jr, MD, Principal Investigator — Lehigh Valley Hospital
Locations (1):
- Lehigh Valley Health Network, Allentown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Murphy S., Kane B., Barr G., Rupp V., Fredericks K., Barraco R., Anselmo T., Reed J., The Correlation Between Adolescent-Reported Parental Driving Behaviors and Observed Adult Driving Behaviors. Annals of Emergency Medicine 54(3):s126-s127, 2009